CLINICAL TRIAL: NCT05850741
Title: Prospective Cardiac Ultrasound Imaging Study With Demonstrator
Acronym: CARDIOKIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Roberto Rordorf, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRCCSSanMatteoPavia
Record Dates: First submitted 2023-04-29; First posted 2023-05-09 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Ventricular Tachycardia
Keywords: artificial intelligence; cardiac radioablation; echocardiography; motion monitoring; ventricular arrhythmia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device (Experimental): The following procedure steps will take place:
  * The study system is installed in the room before patient arrival
  * The patient needs to fully undress the upper body before lying on the bed
  * The 3 ECG electrodes are placed
  * Ultrasound gel is applied on the ultrasound probe
  Interventions: Device: Cardiokit

INTERVENTIONS:
Device: Cardiokit — The CardioKit prototype used in the study can monitor cyclical heart-beat motion, cyclical respiratory motion and non-cyclical heart position changes while the patient is lying in supine position.

SUMMARY:
The Prospective Cardiac Ultrasound Imaging Study is a single center, single arm, feasibility study. The study aims at collecting cardiac ultrasound data from patients diagnosed with ventricular tachycardia, during rest and short breath hold sequences. This study is part of the engineering studies linked to the CardioKit-Minimum Viable Product project. The CardioKit prototype used in the study can monitor cyclical heart-beat motion, cyclical respiratory motion and non-cyclical heart position changes while the patient is lying in supine position.

DETAILED DESCRIPTION:
The research will analyse the ultrasound image data quality, especially investigating the ability of the prototype system to automatically and correctly interpret ultrasound images and artifact issues which may arise from age, body composition, mechanical valves, leads from implanted devices, or other implants. The study will establish if it is appropriate to develop a new medical device supporting automated cardiac ultrasound image interpretation during non-invasive cardiac procedures, i.e. ventricular tachycardia stereotactic radioablation. This early research protocol did collect data from 24 adult patients. The data were not used for diagnostic nor treatment purposes and the protocol's procedure duration was limited to one hour, hence the research was considered of very limited risk for the participants. The research will provide a Proof-of-Concept for a Medical Device to benefit patients with ventricular tachycardia and other cardiac pathologies in the future.

ELIGIBILITY:
Inclusion criteria:

1. Patient with history of ventricular tachycardia
2. Over 18 years old
3. Ability and willingness to provide written informed consent

Exclusion criteria:

1. Patient in arrhythmic storm

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
Image quality in terms of allowing a correct identification of the phase of the cardiac cycle by the prototype software. | Baseline
  The primary endpoint was defined as the percentage of patients able to obtain a positive result in a multi parametric score of image quality, consisting of:
  Score = 1: average phase error per patient, defined as the difference between the phase of the cardiac cycle identified by the algorithm and the one evaluated by the ECG reference <0.1.
  Score = 0: average phase error per patient ≥0.1.
  For each patient, scoring was done for each imaging view (i.e., parasternal and apical). If the score was 2 (at least 1 point in A or B and 1 point in C or D) or greater for at least one of the imaging views, the outcome was considered as positive. The final result is the proportion of patients (in %) with a positive outcome, defined as the number of patients with a positive evaluation divided by the total number of patients x 100.
Image quality in terms of allowing a correct measurement of the heart displacement (mainly due to respiratory motion) by the prototype software. | Baseline
  The primary endpoint was defined as the percentage of patients able to obtain a positive result in a multi parametric score of image quality, consisting of:
  Score = 1: maximum excursion calculated by the algorithm <30 mm with a total 3D error in the calculation of the displacement <3 mm.
  Score = 0: either maximum excursion calculated by the algorithm ≥30 mm or total 3D error in the calculation of the displacement ≥3 mm (or both).
  For each patient, scoring was done for each imaging view (i.e., parasternal and apical). If the score was 2 (at least 1 point in A or B and 1 point in C or D) or greater for at least one of the imaging views, the outcome was considered as positive. The final result is the proportion of patients (in %) with a positive outcome, defined as the number of patients with a positive evaluation divided by the total number of patients x 100.
Image quality in terms of the ability to distinguish typical cardiac structures, as assessed visually by the clinical operator. | Baseline
  The primary endpoint was defined as the percentage of patients able to obtain a positive result in a multi parametric score of image quality, consisting of:
  Score = 1: ability to identify visually by an experienced operator in the acquired image at least one of the following structures: left ventricular free wall, interventricular septum, mitral valve, or aortic valve.
  Score = 0: inability to identify at least one of these structures.
  For each patient, scoring was done for each imaging view (i.e., parasternal and apical). If the score was 2 (at least 1 point in A or B and 1 point in C or D) or greater for at least one of the imaging views, the outcome was considered as positive. The final result is the proportion of patients (in %) with a positive outcome, defined as the number of patients with a positive evaluation divided by the total number of patients x 100.
Image quality in terms of the stability of the image throughout the respiration cycle, as assessed visually by the clinical operator. | Baseline
  The primary endpoint was defined as the percentage of patients able to obtain a positive result in a multi parametric score of image quality, consisting of:
  Score = 1: persistence of cardiac structures within the echocardiographic image during respiratory motion.
  Score = 0: disappearance of cardiac structures from the echocardiographic image during respiratory motion.
  For each patient, scoring was done for each imaging view (i.e., parasternal and apical). If the score was 2 (at least 1 point in A or B and 1 point in C or D) or greater for at least one of the imaging views, the outcome was considered as positive. The final result is the proportion of patients (in %) with a positive outcome, defined as the number of patients with a positive evaluation divided by the total number of patients x 100.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Rordorf, md, Principal Investigator — Fondazione IRCCS Policlinico San Matteo di Pavia
Locations (1):
- IRCCS Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/41/NCT05850741/Prot_000.pdf